CLINICAL TRIAL: NCT04016103
Title: MY01 - An Aid for Diagnosing Acute Compartment Syndrome in Real Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MY01 Inc. (Industry)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MY01 - QC - 01
Record Dates: First submitted 2019-07-03; First posted 2019-07-11 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Acute Compartment Syndrome
Keywords: Acute Compartment Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MY01 Device (Experimental): Insertion of the MY01 device for up to 24 hours for continuous monitoring of compartment pressure
  Interventions: Device: MY01 - Continuous Compartmental Pressure Monitor

INTERVENTIONS:
Device: MY01 - Continuous Compartmental Pressure Monitor — Insertion of the MY01 device for up to 24 hours for continuous monitoring of compartment pressure

SUMMARY:
Compartment syndrome can result from extremity trauma. It can also be caused by procedural cases that involve lower or upper extremity surgery. This condition results in muscle death, chronic pain, infection, and possible amputation. Early diagnosis is essential to institute interventions that can avoid complications. Subjective pain of the patient remains the mainstay for diagnosis. A method or device is needed that would improve our accuracy in diagnosing compartment syndrome. Ideally, this would be suited for single and/or continuous pressure read-outs. The aim is to reduce the incidence of missed compartment syndrome and diminish delays that would lead to significant disability.

Despite awareness, delayed diagnosis and treatment occurs in modern orthopaedic practice. As noted in many studies, once a diagnosis has been made, immediate fasciotomy is necessary to provide the best chance for a favourable clinical result. Therefore, there is a need for improved devices in order to obtain an early and reliable diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged 18 years of age and older
* Any tibial, foot, femoral, forearm or fracture that is felt by the surgeon to have a reasonable indication that elevated ICP could occur in the patient
* Mentally fit to provide informed consent

Exclusion Criteria:

* Patients with fractures that are not felt to be at risk of developing compartment syndrome based on serial clinical evaluation
* Infected wounds; infected fractures
* Patients who present with ACS requiring urgent surgical fasciotomy
* Patients who cannot consent to trial
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical ease with which the new compartment pressure monitor was inserted into compartment. | 24-48 hours following device insertion
  At device insertion, the physician will complete a feedback questionnaire, and routine assessment will be performed in compliance with the standard of care. As part of the feedback questionnaire, the physician will be asked to indicate on a sliding scale "How certain are you the device functioned adequately?" [0 = not confident] - [10 = very confident].
  The scale, administered part of a Clinical Report Form (CRF) titled 'Physician Survey', measures the physicians subjective level of certainty that the device sensor was inserted correctly within a patients muscle compartment. A record of 10 should be considered a very positive scenario, whereas a record of 0 should indicate a very negative scenario.
Ability to monitor in real-time the continuous pressure read-out from the compartment in remote locations such as an I-phone. | 24-48 hours following device insertion
  At device insertion, the physician will complete a feedback questionnaire, and routine assessment will be performed in compliance with the standard of care. As part of the feedback questionnaire, the physician will be asked to indicate in a Yes or No question "Did the MY01 Application remote data display work properly?" [Yes] or [No].
The correlation of continuous pressure read-outs (high, normal or low) with clinical indications for compartment syndrome in each patient. | 24-48 hours following device insertion, and again during the final follow-up of the participant approximately two weeks after treatment
  Routine assessments will be completed by healthcare personnel as per standard of care (the 6P's [Pain, Paraesthesia, Pallor, Paralysis, Pulselessness, Poikilothermia]), and compared against the pressure readout [mmHG] indicated by MY01's MicroElectroMechanical (MEMS) pressure sensor inserted at the afflicted location.

SECONDARY OUTCOMES:
Correlation of clinical compartment syndrome release with data from the continuous pressure monitor read-out. | 24-48 hours following device insertion, and again during the final follow-up of the participant approximately two weeks after treatment
  Should surgical fasciotomy be deemed necessary to release pent up pressure in the patients muscle compartment, the continuous pressure read-outs [mmHG] derived from the device will be compared against the timeframe when the decision to conduct fasciotomy was made.
Short-term outcomes of the patient following continuous pressure monitoring | 24-48 hours following device insertion.
  Survey and tabulation of data from patient clinical findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Bernstein, MD, Principal Investigator — Staff Surgeon, Orthopaedic Trauma & Limb Deformity, Montreal General Hospital | Assistant Professor Department of Surgery and Pediatric Surgery McGill University
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No